CLINICAL TRIAL: NCT01168869
Title: Myocardial Infarction as the First Manifestation of Coronary Heart Disease: Rates of Heralded and Unheralded Myocardial Infarction. A CALIBER Study
Brief Title: Myocardial Infarction as the First Manifestation of Coronary Heart Disease: Rates of Heralded and Unheralded Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: British Medical Research Council (Other Government); University College, London (Other)
Responsible Party: Principal Investigator, Emily Herrett, Dr, London School of Hygiene and Tropical Medicine
Other Study IDs: CALIBER 09-07; 086091/Z/08/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2010-07-19; First posted 2010-07-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Infarction
Keywords: Manifestation; Coronary Heart Disease; Myocardial infarction; Angina pectoris; Unheralded; General Practice Research Database; Myocardial Ischaemia National Audit Project; CALIBER
MeSH Terms: conditions — Myocardial Infarction; Coronary Disease; Angina Pectoris

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GPRD patients: All patients included in "up to standard" GPRD practices that agreed to the linkage with the MINAP database are included in this cohort.

SUMMARY:
Some myocardial infarctions (MI) occur as the first manifestation of coronary artery disease. These are termed 'unheralded' events as they have not been preceded by other forms of coronary artery disease. Unheralded MIs are important because of the high likelihood of missed opportunities for prevention. The proportion of MIs that are 'unheralded' is unknown.

This study aims to quantify the proportion of MIs that occur 'unheralded' and also give an estimate of the incidence of 'unheralded' MI in the UK, compared to 'heralded' MI and those with angina of recent onset (MIs with premonitory symptoms).

DETAILED DESCRIPTION:
This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

Using data from MINAP and GPRD, patients experiencing their first myocardial infarction (MI) will be separated into three categories:

* 'Heralded MI': patients who have been diagnosed or treated for cardiovascular disease for more than 90 days before MI.
* 'MI with premonitory symptoms': patients who have been diagnosed or treated for cardiovascular disease within the 90 days prior to MI.
* 'Unheralded MI': patients without a cardiovascular disease diagnosis or treatment at any time before MI.

Patients with MI will be identified in the linked GPRD-MINAP record. Using GPRD population denominators, this study will establish the absolute incidence rates of first 'unheralded' MI by calendar year, age, sex, season, MI subtype (ST-elevation MI and non ST-elevation MI) and region and compare these to the rates of first 'heralded' MIs and first 'MI with premonitory symptoms'.

ELIGIBILITY:
Inclusion Criteria:

* Patients in GPRD practices which are deemed "up to standard" by GPRD criteria will be included if their practice agreed to be linked to the MINAP dataset.
* Age over 18.

Exclusion Criteria:

* Patients will be excluded after experiencing their first MI.
* Patients will be excluded if they do not fulfil one of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients registered at those GPRD practices that agreed to the linkage with the MINAP database, and whose practices are "up to standard" according to GPRD criteria. Practices taking part in the GPRD are chosen to be representative of all UK practices, and 98% of people in the UK are registered with a GP. Therefore the GPRD should be a representative sample of the UK population.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
First myocardial infarction (MI) | Average time frame: patients in the GPRD are followed from registration until they experience the outcome, leave the practice, die, or 31st December 2009, whichever occurs first.
  First MIs will be divided into three groups:
  (i) Those with previous manifestations of cardiovascular disease, diagnosed or treated more than 90 days before the MI. These are the 'Heralded MIs'.
  (ii) Those with a diagnosis or treatment of cardiovascular disease occurring only within 90 days before MI. These are the 'MIs with premonitory symptoms'.
  (iii) Those without any previous manifestation of cardiovascular disease at any time before MI. These are the 'Unheralded MIs'.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Herrett, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Harry Hemingway, FRCP, Study Director — University College, London
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom